CLINICAL TRIAL: NCT04923620
Title: Efficacy and Safety of Neoadjuvant Cetuximab + Chemotherapy Combined With Short-course Radiotherapy for RAS Wild-type Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Cetuximab + Chemotherapy Combined With Short-course Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Principal Investigator, Cai Zhenghao, MD, Shanghai Minimally Invasive Surgery Center
Other Study IDs: MISC-Cet-FOLFOX-SCRT
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Neoadjuvant Treatment; Rectal Cancer; Cetuximab; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cetuximab+mFOLFOX6 — cetuximab 500mg/m2 d1 Oxaliplatin 85mg/m2 d1 Calcium Folinate 400mg/m2 d1 5-fluorouridine 400mg/m2 d1 5-fluorouridine 2400mg/m2 46h q2w, 6 cycles
Radiation: short-course radiotherapy — 25Gy/5Fx short-course radiotherapy between the forth and the fifth cycle of cetuximab+mFOLFOX6

SUMMARY:
Prospectively Investigate the effectiveness and safety of neoadjuvant cetuximab + chemotherapy (mFOLFOX6) combined with short-course radiotherapy (25Gy/5Fx) for RAS wild-type locally advanced rectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. A biopsy proven histological diagnosis of rectal adenocarcinoma；
2. An ARMS-PCR proven KRAS, NRAS, PI3KCA and BRAF wild type;
3. No intestinal obstruction, distant metastasis was excluded by CT, MRI or PET / CT;
4. MRI proven T3c-T4, CRM positive, N2, extramural vascular invasion positive or lateral lymph node positive of locally advanced rectal cancer;
5. Age between 18-75 years;
6. ECOG (Eastern US Cooperative Oncology Group) score: 0-1;
7. Has sufficient organ function:

   * Hemopoietic function: hemoglobin ≥ 90 g / L, platelet ≥ 80 g / L × 109 / L, neutrophils ≥ 1.5 × 109/L
   * Liver function: ALT and AST < 2.5 × ULN;
   * Renal function: serum creatinine < 1.5 ULN;
8. Willing to participate and informed consent signed；

Exclusion Criteria:

1. Patients with mutations in any of KRAS, NRAS, or BRAF, microsatellite instablility-High;
2. Patients having undergone chemotherapy, radiotherapy or surgery for colorectal cancer;
3. Patients with other uncontrolled malignant tumors (except early-stage basal cell carcinoma or cervical carcinoma in situ) ;
4. Female patients who are pregnant or breastfeeding;
5. Patients with severe heart, liver, or kidney, or neurological or psychiatric disease;
6. Patients with active infection;
7. Poor overall health status, ECOG ≥ 2;
8. Patients with concomitant diseases that seriously endanger the safety of patients or affect the completion of the study in the judgment of the investigator;
9. Known hypersensitivity reactions to any investigational drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 75 years with locally advanced rectal cancer, regardless of gender, ethnicity and regional distribution, were involved in this study. Patients were required to be in good health and have sufficient organ function and bone marrow function.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | two weeks after surgery
  Tumor Regression Grade 0-1

SECONDARY OUTCOMES:
Pathological complete response rate | two weeks after surgery
  Refers to the pathological examination of primary tumors and lymph node surgical specimens without residual infiltrating tumor cells (ypT0N0, TRG 0)
2-year local control rate | 2 years after enrollment
  Refers to the probability of not finding local recurrence of tumor within 2 years，including anastomotic recurrence confirmed by pathological biopsy, pelvic tumor recurrence confirmed by imaging examination, or suspected pelvic recurrence with CEA exceeding the normal upper limit.
2-year metastasis-free rate 2-year distant metastasis free rate | 2 years after enrollment
  Refers to the probability of no distant metastasis within 2 years
Overall survival | 2 years after enrollment
  Refers to the time from the start of treatment to death due to any cause.
disease-free survival | 2 years after enrollment
  Refers to the time from the start of treatment to recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China